CLINICAL TRIAL: NCT05254912
Title: Evaluation of Topically Applied Bemotrizinol for Human Photoallergic Potential
Brief Title: Photoallergic Potential of 6% Bemotrizinol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DSM PA 2020
Record Dates: First submitted 2022-02-11; First posted 2022-02-24 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Photoallergic Response
Keywords: Sunscreen, photoprotective, UV-filter
MeSH Terms: interventions — bis-ethylhexyloxyphenol methoxyphenyl triazine; Petrolatum

STUDY DESIGN:
Intervention Model Description: This study will evaluate the potential of an investigational product (6% Bemotrizinol (BEMT) in a suitable vehicle (i.e., sunscreen oil SU E 101413 85) or petrolatum (SU-E-101413-82)) to produce a photoallergic response after application to the skin of human subjects followed by exposure to UV radiation.
Who Masked: Participant
Masking Description: Subjects will be blinded to the name of the investigational products. The Investigatory staff will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 6% BEMT in sunscreen oil (SU E 101413 85) (Active Comparator): Assess the photoallergic potential of Sunscreen oil with 6% BEMT (PARSOL® Shield) and 10% ethanol as penetration enhancer a test material (formulation: SU E 101413 85).
  Approximately 0.15 g or 0.15 ml of each product and vehicle control will be applied. Two doses (one irradiated and one non- irradiated) of the investigational products and two doses (one irradiated and one non- irradiated) of the vehicle controls will be applied to back of each subject once on Day 1 under occlusive patches. Patches will remain in place for approximately 24 hours and will be removed by clinical study staff on Day 2. During the challenge phase, two undosed negative control occlusive patches will also be also applied. Subjects will return to the laboratory 24 hours and 48 hours post-irradiation for dermal evaluations. Dermal scores obtained during the challenge phase will be reported for each site.
  Interventions: Drug: 6% Bemotrizinol in sunscreen formulation
- Sunscreen oil Vehicle (SU E 101413 91) (Other): Vehicle Control: Assess the photoallergenic potential of sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT.
  Approximately 0.15 g or 0.15 ml of each product and vehicle control will be applied. Two doses (one irradiated and one non- irradiated) of the investigational products and two doses (one irradiated and one non- irradiated) of the vehicle controls will be applied to back of each subject once on Day 1 under occlusive patches. Patches will remain in place for approximately 24 hours and will be removed by clinical study staff on Day 2. During the challenge phase, two undosed negative control occlusive patches will also be also applied. Subjects will return to the laboratory 24 hours and 48 hours post-irradiation for dermal evaluations. Dermal scores obtained during the challenge phase will be reported for each site.
  Interventions: Other: Vehicle
- 6% BEMT in petrolatum (SU E 101413 82) (Active Comparator): Assess the photoallergenic potential of a dispersion of 6% BEMT (PARSOL® Shield) in petrolatum
  Approximately 0.15 g or 0.15 ml of each product and vehicle control will be applied. Two doses (one irradiated and one non- irradiated) of the investigational products and two doses (one irradiated and one non- irradiated) of the vehicle controls will be applied to back of each subject once on Day 1 under occlusive patches. Patches will remain in place for approximately 24 hours and will be removed by clinical study staff on Day 2. During the challenge phase, two undosed negative control occlusive patches will also be also applied. Subjects will return to the laboratory 24 hours and 48 hours post-irradiation for dermal evaluations. Dermal scores obtained during the challenge phase will be reported for each site.
  Interventions: Drug: 6% Bemotrizinol in petrolatum

INTERVENTIONS:
Drug: 6% Bemotrizinol in sunscreen formulation — 6% Bemotrizinol (BEMT) in a basic sunscreen oil formulation (SU E 101413 85)
  Other Names: PARSOL SHIELD
  Arms: 6% BEMT in sunscreen oil (SU E 101413 85)
Drug: 6% Bemotrizinol in petrolatum — 6% Bemotrizinol (BEMT) as a dispersion in petrolatum (SU-E-101413-82)
  Other Names: PARSOL SHIELD
  Arms: 6% BEMT in petrolatum (SU E 101413 82)
Other: Vehicle — Sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT (SU E 101413 91)
  Arms: Sunscreen oil Vehicle (SU E 101413 91)

SUMMARY:
This clinical trial will assess the photoallergic potential of BEMT (6%), compared to a vehicle control and a negative control.

DETAILED DESCRIPTION:
The primary endpoint of this clinical trial is to evaluate the potential of Bemotrizinol (6%) to produce a photoallergic response.

The potential of 6% Bemotrizinol to produce a photoallergic response after application to the skin of human subjects followed by exposure to ultraviolet (UV) radiation will be assessed via the evaluation of a sunscreen oil with 6% BEMT and 10% ethanol as penetration enhancer (SU E 101413 85), as compared to a sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT (SU-E-101413-82) and a dispersion of 6% BEMT in petrolatum (SU-E-101413-82).

Upon enrollment, a site on a subject's lower back, isolated from the actual test site, will be chosen to determine the subject's Minimal Erythema Dose (MED). The MED of each subject is assessed by applying a progressive geometric sequence of UV radiation exposures to five sub-sites, each of which is graduated incrementally by 25% over the previous site. The MED is evaluated 16 to 24 hours after ultraviolet radiation.

Duplicate test sites on the back (each approximately 4 cm2) will be identified. Test material will be applied to designated patches and affixed to both sides of the back. One side will be designated for irradiation, and the other is used as a treated/non-irradiated control. Approximately 0.15 g of each investigational product or vehicle controls will be applied to the fabric portion of separate patches with occlusive strips; an un-dosed patch will also be used.

Approximately 24 hours after application, the patches will be removed and the skin will be gently wiped. The MED will be determined from the five UV-treated sub-sites and all of the test sites will be evaluated according to the erythema grading scale. The sites designated for irradiation will be then irradiated with solar simulated light by two times an individual's MED.

The remaining site serves as the non-irradiated control. Test sites are delineated with a marking pen to ensure continuity of patch application and patch site location.

There will be three study phases associated with this study: Induction, challenge and re-challenge.

The induction phase procedure will be carried out twice weekly for a total of six applications/post-irradiation readings. However, the schedule may be modified to accommodate inclement weather, holidays, or missed applications. At the discretion of the Principal Investigator, the test material may then be applied, the sites irradiated and scored on two consecutive days during the Induction Phase. If a patch and or irradiation is missed, a 3-day sequence of patch/irradiation/score will be added at the end of the Induction Phase. Subjects must have no fewer than 5 evaluations at the end of the Induction phase. Only one rescheduled patch or irradiation procedure is permitted. Subjects missing a second visit are discontinued from the study due to non-compliance with the study protocol. For evaluation of photoallergy, during the Induction Phase, the sites are irradiated with 2 times the subject's MED (full spectrum wavelengths UVB 290-320 nm and UVA 320-400 nm) J/cm2 UVA. During the challenge phase, the sites will be irradiated with a dose of 10 J/cm2 of UVA light (320-400 nm) using cut-off filters to block UVB wavelength 290-320 nanometers.

Irradiated area within the treated sites and control sites are examined approximately 24 hours following irradiation of the test sites and graded. Skin condition of the sites will be evaluated at each visit for possible skin reactions to the test material. Any reaction will be documented on the source document.

If a 2+ reaction or greater occurs on a site, the application of the test material may be discontinued for the remainder of the Induction Phase, but may be challenged on the appropriate day of the study.

At the discretion of the Principal Investigator, subjects exhibiting a significant reaction at the beginning of the Induction Phase may be considered to be "pre-sensitized" to an ingredient(s) of the test product and may be discontinued from the patching and irradiation of that test material for the remainder of the study.

The challenge phase will occur approximately 10 to 21 days following the last induction application. Duplicate patches are applied to sites previously unexposed to the test material. In addition, 2 sets of patches without test material will be also applied on 2 sides of the back. Approximately 24 hours later, the patches are removed, the test sites are evaluated. The test sites on one side of the back are irradiated with a non-erythrogenic dose of Ultra Violet A (UVA) radiation (wavelengths 320-400 nm) equivalent to approximately 10 J/cm². The sites on the other side of the back serve as a "test material treated, non-irradiated" control site and "non-treated, non-irradiated" control. The challenge sites are graded at 24, 48, and 72 hours following irradiation according to the dermal grading scale.

A re-challenge phase may be initiated at the discretion of the Investigator, and with the Sponsor's approval. A subject may be re-challenged with the test material if reactions indicative of sensitization or photo sensitization are observed during the Challenge Phase. The subject(s) will be asked to return to the laboratory no sooner than two weeks following the conclusion of the PA study and the Challenge procedures will be repeated. One patch of the test material will be applied to the subject's back and allowed to remain in direct contact with the skin for 24 hours. The subject will return after 24 hours for removal of the patch and grading of the site, without irradiation if sensitization is suspected or with irradiation of an additional treated site (24 hour exposure) if reactions suggestive of photosensitization are observed during the study. Subjects will return for a 48 hour and 72 hour post-patch application grading and additional 96 hour evaluation if a reaction persists. If the sites are irradiated after patch removal, subjects will return for evaluation at 24 hour, 48 hour and 72 hour post UV exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between 18 and 75 years of age;
2. Subject has a Fitzpatrick Skin Types I - III, based on the first 30 to 45 minutes of sun exposure after a winter season of no sun exposure according to the following criteria; I Always burns easily; never tans (sensitive) II Always burns easily; tans minimally (sensitive) III Burns moderately; tans gradually (normal)
3. Subject agrees to avoid excessive sun exposure of the test sites and to refrain from visits to tanning salons during the course of this study;
4. Subject does not exhibit any skin diseases or abnormalities which might be confused with a skin reaction from the test material;
5. Subject agrees not to introduce any new cosmetic or toiletry products during the study;
6. Subject agrees to refrain from getting patches wet and from scrubbing or washing the test area with soap or applying powders, lotions or personal care products to the area during the course of the study;
7. Subject is dependable and able to follow directions as outlined in the protocol and anticipates being available for all study visits;
8. Subject is willing to participate in all study evaluations;
9. Subject is in generally good health and has a current Panelist Profile Form on file at CRL;
10. Subject has completed a HIPAA Authorization Form in conformance with 45 CFR Parts 160 and 164;
11. Subject understands and is willing to sign an Informed Consent Form in conformance with 21 CFR Part 50: "Protection of Human Subjects."

Exclusion Criteria:

1. Female subject is pregnant, nursing, planning a pregnancy, or not using adequate birth control;
2. Subjects with a prior history of phototoxic or photoallergic reactions or those taking medication which might produce an abnormal response to sunlight;
3. Subject has received treatment with sympathomimetics, antihistamines, vasoconstrictors, non-steroidal anti-inflammatory agents, and/or systemic or topical corticosteroids within one week prior to initiation of the study;
4. Subject has a history of acute or chronic dermatologic, medical, and/or physical conditions which would preclude application of the test material and/or could influence the outcome of the study;
5. Subject is under treatment for a skin and/or systemic bacterial infection;
6. Subject reports a history of allergies to tape adhesives;
7. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study;
8. Subject has known allergies to sunscreen, skin treatment products or cosmetics, toiletries, and/or topical drugs;
9. Subject has a known communicable disease (e.g., HIV, sexually transmitted diseases, Hepatitis B, Hepatitis C, etc.);
10. Subject has insulin-dependent diabetes;
11. Subject has a history of cancer;
12. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study;
13. Subject exhibits sunburn, suntan, uneven skin tone, blemishes, moles or excess hair in the test site area.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Photoallergy potential of a BEMT (6%) formulation based on a dermal scoring system 24 hours post irradiation | Photoallergy response will be evaluated 24 hours post irradiation
  Photoallergenicity conclusions (i.e., "Photoallergic Response" or "Not a contact sensitizer or photoallergen") will based on a comparison of the reactions obtained on treated/irradiated, treated/non-irradiated and non- treated control sites. Investigational product safety will be determined through interpretation of the dermal evaluation scores.
  The following dermal scoring system will be used to evaluate the irradiated area within the treated test site:
  Grading scale for Erythema:
  "0" = No visible skin reaction; "+" = Barely perceptible erythema; "1+" = Mild erythema; "2+" = Well defined erythema; "3+" = Severe erythema
  Grading Scale for dermal response:
  e = Edema P = Peeling S = Spreading of reaction beyond irradiated site. Sc = Scabbing d = Dryness/scaling D = Oozing, crusting, and/or superficial erosions I = Itching Pa = Papules V = Vesicle W = Weeping Hr = Hyperpigmentation Ho = Hypopigmentation M = Missed Visit
Photoallergy potential of a BEMT (6%) formulation based on a dermal scoring system 48 hours post irradiation | Photoallergy response will be evaluated at 48 hours post irradiation
  Photoallergenicity conclusions (i.e., "Photoallergic Response" or "Not a contact sensitizer or photoallergen") will based on a comparison of the reactions obtained on treated/irradiated, treated/non-irradiated and non- treated control sites. Investigational product safety will be determined through interpretation of the dermal evaluation scores.
  The following dermal scoring system will be used to evaluate the irradiated area within the treated test site:
  Grading scale for Erythema:
  "0" = No visible skin reaction; "+" = Barely perceptible erythema; "1+" = Mild erythema; "2+" = Well defined erythema; "3+" = Severe erythema
  Grading Scale for dermal response:
  e = Edema P = Peeling S = Spreading of reaction beyond irradiated site. Sc = Scabbing d = Dryness/scaling D = Oozing, crusting, and/or superficial erosions I = Itching Pa = Papules V = Vesicle W = Weeping Hr = Hyperpigmentation Ho = Hypopigmentation M = Missed Visit
Photoallergy potential of a BEMT (6%) formulation based on a dermal scoring system 72 hours post irradiation | Photoallergy response will be evaluated at 72 hours post irradiation
  Photoallergenicity conclusions (i.e., "Photoallergic Response" or "Not a contact sensitizer or photoallergen") will based on a comparison of the reactions obtained on treated/irradiated, treated/non-irradiated and non- treated control sites. Investigational product safety will be determined through interpretation of the dermal evaluation scores.
  The following dermal scoring system will be used to evaluate the irradiated area within the treated test site:
  Grading scale for Erythema:
  "0" = No visible skin reaction; "+" = Barely perceptible erythema; "1+" = Mild erythema; "2+" = Well defined erythema; "3+" = Severe erythema
  Grading Scale for dermal response:
  e = Edema P = Peeling S = Spreading of reaction beyond irradiated site. Sc = Scabbing d = Dryness/scaling D = Oozing, crusting, and/or superficial erosions I = Itching Pa = Papules V = Vesicle W = Weeping Hr = Hyperpigmentation Ho = Hypopigmentation M = Missed Visit

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Schutz, PhD, Study Director — DSM Nutritional Products, Inc.; Gladys Osis, MT, Principal Investigator — Eurofins CRL Inc.
Locations (1):
- Eurofins | CRL, Inc., Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No